CLINICAL TRIAL: NCT05910333
Title: Ten Years Retrospective Study of 4 LOCATOR Attachment of Mandibular Implant Retained Overdenture With 2 Different Distributions.
Brief Title: Four Locator Attachment Mandibular Overdentures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mohamed Elsawy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Elsawy, lecturer, Department of prosthodontics, principle investigator, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: A0103023RP
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quadrilateral distribution group: Patients with quadrilateral distribution of implants
  Interventions: Other: observation
- Linear distribution group: Patients with lineardistribution of implants
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — To compare the effect of the mandibular implant retained OVD using quadrilateral distribution (QD) versus linear distribution (LD) on posterior mandibular ridge resorption (PMandRR), anterior maxillary ridge resorption (AMaxRR), and changes to the crestal bone level around implants after 10 years of function.

SUMMARY:
. There is little information on the degree of crestal bone loss around 4 inter-foraminal implant-retained mandibular overdentures (OVDs) and the amount of bone remodelling on the anterior maxilla and posterior mandibule on long-term function, particularly with different distributions.

DETAILED DESCRIPTION:
Numerous studies confirm the successful use of implants to retain prostheses in the edentulous atrophic mandible. It has been recommended by some authors that clinicians should use 3 or 4 implants in situations that require increased retention, such as high muscle attachment or prominent mylohyoid ridge. LOCATOR attachment as a retentive component has several advantages over other systems, Such as: dual retention through both external and internal mating surfaces, a self-aligning feature which is helpful in guiding patients when placing their denture. There is little information on the degree of crestal bone loss around 4 inter-foraminal implant-retained mandibular overdentures (OVDs) and the amount of bone remodelling on the anterior maxilla and posterior mandibule on long-term function, particularly with different distributions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 4 implants in the inter-foraminal region.
* Patients treated by staff and students in the Master's program in Prosthodontics Department according to the following criteria:
* Edentulous maxilla and mandible for at least 1 year.
* Problems with retention and stability of the mandibular denture.
* Mandibular bone height between 15 and 25 mm.

Exclusion Criteria:

* Patients with relative contraindications, such as
* A history of para functional habits.
* Smokers more than 10 cigarettes per day.
* alcoholism.
* Patients with a history of radiation therapy in the head and neck region . • Patients within intravenous administrated bisphosphonates., chemotherapy, and mental disorders that could jeopardies their co-operation.

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — above 60
Study Population: 10 patients in each group. total number of patients 20.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-10-21 (Estimated); Study Completion 2023-10-27 (Estimated)

PRIMARY OUTCOMES:
Posterior mandibular ridge resorption (PMandRR) | 10 years retrospective study
  The amount of PMandRR will be assessed using posterior area index on a panoramic x-ray which use specific landmarkds.

SECONDARY OUTCOMES:
Anterior maxillary ridge resorption (AMaxRR) | 10 years
  The amount of PMandRR will be assessed using anterior area index on a panoramic x-ray, which use specific landmarks.

OTHER OUTCOMES:
Crestal bone loss around implants | 10 years
  amount of bone loss which appears on a periapical radiograph.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Sawy, Study Director — Mansoura University
Locations (1):
- Mohammed El Sawy, Multiple Locations, Egypt

IPD SHARING:
Plan to Share IPD: No
just by contacting the corresponding author